CLINICAL TRIAL: NCT06689124
Title: A Randomized Study Comparing of Three Doses Nebulized Fentanyl in Older Adults with Severe Musculoskeletal Pain At the Emergency Department
Brief Title: A Randomized Study Comparing of Three Doses Nebulized Fentanyl in Older Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bangkok Metropolitan Administration Medical College and Vajira Hospital (Other Government)
Collaborators: Navamindradhiraj University (Other)
Responsible Party: Principal Investigator, Thananda Trakarnvanich, Doctor, Bangkok Metropolitan Administration Medical College and Vajira Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 219/66 FB
Record Dates: First submitted 2024-06-04; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Treatment Side Effects; Musculoskeletal Pain
Keywords: fentanyl; opioid; nebulized; musculoskeletal pain; elderly; emergency room; randomized controlled trial; Thai
MeSH Terms: conditions — Musculoskeletal Pain; Emergencies

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Nebulized fentanyl 2 mcg/kg (Active Comparator): The researcher prepared fentanyl (the researcher informed the in-charge nurse to open the medicine cabinet and double-checked the dosage with the in-charge nurse). The dosage was 2 micrograms per kilogram of body weight (calculated based on the patient's actual weight in kilograms). The medication was contained in a nebulizer. It was then mixed with normal saline (0.9% normal saline) to a total volume of 5 milliliters and administered via nebulization.
  Interventions: Drug: Nebulized fentanyl
- Nebulized fentanyl 3 mcg/kg (Active Comparator): The researcher prepared fentanyl (the researcher informed the in-charge nurse to open the medicine cabinet and double-checked the dosage with the in-charge nurse). The dosage was 3 micrograms per kilogram of body weight (calculated based on the patient's actual weight in kilograms). The medication was contained in a nebulizer. It was then mixed with normal saline (0.9% normal saline) to a total volume of 5 milliliters and administered via nebulization.
  Interventions: Drug: Nebulized fentanyl
- Nebulized fentanyl 4 mcg/kg (Active Comparator): The researcher prepared fentanyl (the researcher informed the in-charge nurse to open the medicine cabinet and double-checked the dosage with the in-charge nurse). The dosage was 4 micrograms per kilogram of body weight (calculated based on the patient's actual weight in kilograms). The medication was contained in a nebulizer. It was then mixed with normal saline (0.9% normal saline) to a total volume of 5 milliliters and administered via nebulization.
  Interventions: Drug: Nebulized fentanyl

INTERVENTIONS:
Drug: Nebulized fentanyl — After the enrollment process, the main research assistant will take a brown envelope containing the randomization and hand it to the principal investigator in numerical order. The principal investigator will then open the envelope to determine the group assignment for the patient, revealing which fentanyl nebulization dosage group (2 mcg/kg, 3 mcg/kg and 4 mcg/kg) the patient will be placed in. In this study, participants will be divided into three groups as previously described. We evaluate pain score at 0, 15, 30, 45, 60, 75, 90, 105 and 120 minutes after receiving nebulized fentanyl by a train research assistance who is blind from the treatment dosage.
  Other Names: Nebulized fentanyl dosage

SUMMARY:
This clinical trial compares three different nebulized fentanyl dosages for older persons experiencing severe musculoskeletal pain at the emergency department.

The main objective is:

Does the effectiveness of nebulized fentanyl at dosages of 2 mcg/kg, 3 mcg/kg, and 4 mcg/kg at 30 minutes differ in older patients who report to the emergency room with pain from musculoskeletal injuries?

Secondary outcome are:

1. Incidence of adverse effects after drug administration at minutes 0, 15, 30, 45, 60, 75, 90, 105, 120
2. Incidence of receiving other pain relief treatments (rescue therapy) in minutes 30, 45, 60, 75, 90, 105, 120 Participants will receive an explanation of the study and possible side effects, which may take approximately 5-10 minutes, without affecting the primary treatment of the patients. Consent will be obtained in this study, along with signing or fingerprinting as evidence in the consent form.

DETAILED DESCRIPTION:
Participants will receive nebulized fentanyl for pain reduction at the pre-determined randomized dose, then researchers will follow up assessments of pain levels, vital signs, and any side effects at various intervals.

ELIGIBILITY:
Inclusion Criteria:

* Age more than or equal 65 years old.
* Presented with musculoskeletal pain within 3 days.
* Pain score on verbal numeric rating scale ≥ 5.

Exclusion Criteria:

* Patients need immediate intervention.
* Patients need acute rescue for acute coronary syndrome, respiratory failure, and stroke.
* Creatinine clearance < 30 ml/min, Cirrhosis stage III, IV (present with ascites and varices).
* Trauma >2 organ.
* Comorbidities of chronic obstructive pulmonary disease.
* Take MAO inhibitors within 14 days.
* History of opioid used within 8 hours.
* History of alcohol or drug abuse.
* History of fentanyl allergy.
* Patients with difficulty to communication (e.g. altered mental status, severe dementia (define by 6-items cognitive screening > 12, language barrier).

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy in pain reduction following nebulized fentanyl administration at different dosages. | 30 Minutes
  Efficacy in pain reduction following nebulized fentanyl administration at dosages of 2 mcg/kg, 3 mcg/kg, and 4 mcg/kg in elderly patients presenting to the emergency department with musculoskeletal pain, using verbal numerical rating scale (VNRS) VNRS score ranges from 0 to 10, with a higher score indicating more severe pain. Ten indicates the worst pain, and zero indicates no pain.

SECONDARY OUTCOMES:
Adverse events following nebulized fentanyl administration at different dosages. | 0, 15, 30, 45, 60, 75, 90, 105, 120 Minutes
  Adverse events following nebulized fentanyl administration at dosages of 2 mcg/kg, 3 mcg/kg, and 4 mcg/kg in elderly patients presenting to the emergency department with with musculoskeletal pain
Events of rescue therapy following nebulized fentanyl administration at different dosages. | 30, 45, 60, 75, 90, 105, 120 Minutes
  Events of rescue therapy following nebulized fentanyl administration at dosages of 2 mcg/kg, 3 mcg/kg, and 4 mcg/kg in elderly patients presenting to the emergency department with musculoskeletal pain

CONTACTS AND LOCATIONS:
Overall Officials: Supavit Punyapatipan, M.D., Principal Investigator — Faculty of medicine, Vajira hospital; Jiraporn Sri-on, M.D., Principal Investigator — Faculty of medicine, Vajira hospital
Locations (2):
- Thailand (2):
  - Faculty of Medicine,Vajira Hospital, Bangkok, Bangkok
  - Jiraporn Sri-on, Bangkok, Bangkok

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang HY, Daubresse M, Kruszewski SP, Alexander GC. Prevalence and treatment of pain in EDs in the United States, 2000 to 2010. Am J Emerg Med. 2014 May;32(5):421-31. doi: 10.1016/j.ajem.2014.01.015. Epub 2014 Jan 21. PMID 24560834
- [Background] Chakour MC, Gibson SJ, Bradbeer M, Helme RD. The effect of age on A delta- and C-fibre thermal pain perception. Pain. 1996 Jan;64(1):143-152. doi: 10.1016/0304-3959(95)00102-6. PMID 8867257
- [Background] Asping U, Bagger PV. [Conization of the cervix with a CO2 laser]. Ugeskr Laeger. 1986 Oct 27;148(44):2828-30. No abstract available. Danish. PMID 3097898
- [Background] Pergolizzi J, Boger RH, Budd K, Dahan A, Erdine S, Hans G, Kress HG, Langford R, Likar R, Raffa RB, Sacerdote P. Opioids and the management of chronic severe pain in the elderly: consensus statement of an International Expert Panel with focus on the six clinically most often used World Health Organization Step III opioids (buprenorphine, fentanyl, hydromorphone, methadone, morphine, oxycodone). Pain Pract. 2008 Jul-Aug;8(4):287-313. doi: 10.1111/j.1533-2500.2008.00204.x. Epub 2008 May 23. PMID 18503626
- [Background] Vlaeyen JWS, Linton SJ. Fear-avoidance and its consequences in chronic musculoskeletal pain: a state of the art. Pain. 2000 Apr;85(3):317-332. doi: 10.1016/S0304-3959(99)00242-0. PMID 10781906
- [Background] Teasell R, Dittmer DK. Complications of immobilization and bed rest. Part 2: Other complications. Can Fam Physician. 1993 Jun;39:1440-2, 1445-6. PMID 8324412
- [Background] Tongbua S, Sri-On J, Thong-On K, Paksophis T. Non-inferiority of intranasal ketamine compared to intravenous morphine for musculoskeletal pain relief among older adults in an emergency department: a randomised controlled trial. Age Ageing. 2022 Mar 1;51(3):afac073. doi: 10.1093/ageing/afac073. PMID 35348606
- [Background] Labroo RB, Paine MF, Thummel KE, Kharasch ED. Fentanyl metabolism by human hepatic and intestinal cytochrome P450 3A4: implications for interindividual variability in disposition, efficacy, and drug interactions. Drug Metab Dispos. 1997 Sep;25(9):1072-80. PMID 9311623
- [Background] By the 2023 American Geriatrics Society Beers Criteria(R) Update Expert Panel. American Geriatrics Society 2023 updated AGS Beers Criteria(R) for potentially inappropriate medication use in older adults. J Am Geriatr Soc. 2023 Jul;71(7):2052-2081. doi: 10.1111/jgs.18372. Epub 2023 May 4. PMID 37139824
- [Background] Grape S, Schug SA, Lauer S, Schug BS. Formulations of fentanyl for the management of pain. Drugs. 2010;70(1):57-72. doi: 10.2165/11531740-000000000-00000. PMID 20030425
- [Background] Rosenblum A, Marsch LA, Joseph H, Portenoy RK. Opioids and the treatment of chronic pain: controversies, current status, and future directions. Exp Clin Psychopharmacol. 2008 Oct;16(5):405-16. doi: 10.1037/a0013628. PMID 18837637
- [Background] Farahmand S, Shiralizadeh S, Talebian MT, Bagheri-Hariri S, Arbab M, Basirghafouri H, Saeedi M, Sedaghat M, Mirzababai H. Nebulized fentanyl vs intravenous morphine for ED patients with acute limb pain: a randomized clinical trial. Am J Emerg Med. 2014 Sep;32(9):1011-5. doi: 10.1016/j.ajem.2014.05.051. Epub 2014 Jun 12. PMID 25027194
- [Background] Sabri A, Szalas J, Holmes KS, Labib L, Mussivand T. Failed attempts and improvement strategies in peripheral intravenous catheterization. Biomed Mater Eng. 2013;23(1-2):93-108. doi: 10.3233/BME-120735. PMID 23442240
- [Background] Yalcinli S, Akarca FK, Can O, Sener A, Akbinar C. Factors affecting the first-attempt success rate of intravenous cannulation in older people. J Clin Nurs. 2019 Jun;28(11-12):2206-2213. doi: 10.1111/jocn.14816. Epub 2019 Mar 13. PMID 30786094
- [Background] Puntillo F, Giglio M, Varrassi G. The Routes of Administration for Acute Postoperative Pain Medication. Pain Ther. 2021 Dec;10(2):909-925. doi: 10.1007/s40122-021-00286-5. Epub 2021 Jul 17. PMID 34273095
- [Background] Thompson JP, Thompson DF. Nebulized Fentanyl in Acute Pain: A Systematic Review. Ann Pharmacother. 2016 Oct;50(10):882-91. doi: 10.1177/1060028016659077. Epub 2016 Jul 12. PMID 27413071
- [Background] Hess DR. Nebulizers: principles and performance. Respir Care. 2000 Jun;45(6):609-22. PMID 10894454
- [Background] Bartfield JM, Flint RD, McErlean M, Broderick J. Nebulized fentanyl for relief of abdominal pain. Acad Emerg Med. 2003 Mar;10(3):215-8. doi: 10.1111/j.1553-2712.2003.tb01993.x. PMID 12615585
- [Background] Miner JR, Kletti C, Herold M, Hubbard D, Biros MH. Randomized clinical trial of nebulized fentanyl citrate versus i.v. fentanyl citrate in children presenting to the emergency department with acute pain. Acad Emerg Med. 2007 Oct;14(10):895-8. doi: 10.1197/j.aem.2007.06.036. PMID 17898251
- [Background] Singh AP, Jena SS, Meena RK, Tewari M, Rastogi V. Nebulised fentanyl for post-operative pain relief, a prospective double-blind controlled randomised clinical trial. Indian J Anaesth. 2013 Nov;57(6):583-6. doi: 10.4103/0019-5049.123331. PMID 24403618
- [Background] Moriarty O, McGuire BE, Finn DP. The effect of pain on cognitive function: a review of clinical and preclinical research. Prog Neurobiol. 2011 Mar;93(3):385-404. doi: 10.1016/j.pneurobio.2011.01.002. Epub 2011 Jan 7. PMID 21216272
- [Background] Li L, Liu X, Herr K. Postoperative pain intensity assessment: a comparison of four scales in Chinese adults. Pain Med. 2007 Apr;8(3):223-34. doi: 10.1111/j.1526-4637.2007.00296.x. PMID 17371409
- [Background] Singh V, Gillespie TW, Lane O, Spektor B, Zarrabi AJ, Egan K, Curseen K, Tsvetkova M, Beumer JH, Sniecinski R, Shteamer JW, Switchenko J, Harvey RD. A dose-escalation clinical trial of intranasal ketamine for uncontrolled cancer-related pain. Pharmacotherapy. 2022 Apr;42(4):298-310. doi: 10.1002/phar.2669. Epub 2022 Feb 21. PMID 35146776
- [Background] Imai K, Morita T, Yokomichi N, Mori M, Naito AS, Yamauchi T, Tsukuura H, Uneno Y, Tsuneto S, Inoue S. Association of the RASS Score with Intensity of Symptoms, Discomfort, and Communication Capacity in Terminally Ill Cancer Patients Receiving Palliative Sedation: Is RASS an Appropriate Outcome Measure? Palliat Med Rep. 2022 Apr 8;3(1):47-54. doi: 10.1089/pmr.2021.0087. eCollection 2022. PMID 35558868
- See also: 32. Ding D, Ishag S. Aldrete Scoring System [Internet]. StatPearls; 2023 [cited 2023 Nov 25]. — https://www.ncbi.nlm.nih.gov/books/NBK594237/
- See also: 13. Norman G. Bowery, Fentanyl, Editor(s): S.J. Enna, David B. Bylund, xPharm: The Comprehensive Pharmacology Reference, Elsevier, 2007, Pages 1-5, ISBN 9780080552323 — https://doi.org/10.1016/B978-008055232-3.61745-3